CLINICAL TRIAL: NCT04503369
Title: Observation of Non-technical Skills (e.g. Communication, Team Leader Skills, Teamwork, Situational Awareness Etc.) in the Pre-hospital Care in the Czech Republic
Brief Title: Observation of Non-technical Skills in the Pre-hospital Care in the Czech Republic
Acronym: NTS
Status: Completed | Type: Observational
Sponsor: David Peran (Other Government)
Collaborators: Emergency Medical Services of the Karlovy Vary region, Czech Republic (Unknown); Emergency Medical Services of the Pilsner region, Czech Republic (Unknown)
Responsible Party: Sponsor-Investigator, David Peran, Head of the Education and Training Centre, Emergency Medical Service, Prague
Organization: Emergency Medical Service, Prague (Other Government)
Other Study IDs: ZZSMHP_001_2020
Record Dates: First submitted 2020-07-29; First posted 2020-08-07 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Non-technical Skills
Keywords: non-technical skills; pre-hospital care; emergency medical services; communication; situational awareness; task management; decision making; teamwork; team leading
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EMS crews: Crews of Emergency Medical Services
  Interventions: Behavioral: Non-technical skills

INTERVENTIONS:
Behavioral: Non-technical skills — Teamwork The work of the team consists of information exchange and coordination of all activities performed. In-team communication is always calm and assertive, and team members support each other.
  Task management With the right planning and preparation of individual activities, the likelihood that all standards of care and best practices will be followed increases.
  Situational awareness Situational awareness refers primarily to the collection of information, its understanding and, on that basis, prediction of direction into which the situation will develop. Maintaining situational awareness is crucial in order to move towards the right goal.
  Decision-making With good situational awareness, one is able to keep in mind all information needed to make the correct decision at the right time. In some cases, it is advisable to consult with other team members or to verify their consent to the proposed procedure.
  Communication Communication is a vital tool when working in a team.

SUMMARY:
The aim of the study is to find out if the Emergency Medical Services (EMS) crews are using the non-technical skills (e.g. communication, decision making, situational awareness etc.) in the real practice and how well they use them.

DETAILED DESCRIPTION:
The aim of the study is to find out if the Emergency Medical Services (EMS) crews are using the non-technical skills (teamwork and team leading, communication, decision making, situational awareness and task management) in the real practice and how well they use them. According to the observations of individual crews by field supervisors the use of non-technical skills will be compared between different groups (e.g. resuscitation, trauma, medical problems, non-emergency situations etc.). The comparison between the collaborators of the study is not the subject of the study.

Main hypothesis: The EMS crews are using all of the aspects of non-technical skills appropriately.

The field supervision is also the limitation of the study because it is done by different observers / supervisors, the observation therefore might by affected by subjective feelings. To minimise the subjective view of the situation all of the field supervisors undergo a uniform training of non-technical skills and how to observe and evaluate them.

ELIGIBILITY:
Inclusion Criteria:

* EMS called
* More than 2 crews on the scene
* Field supervisor present

Exclusion Criteria:

- TEAM tool not filled completely

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patient of EMS in participated regions of the Czech Republic where the pre-hospital care is provided by 2 or more crews and the field supervisor is present.
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
NTS incidence | Through study completion, an average of 1 year and until 100 cases from each organization will be collected - 300 observations in total.
  The measurement of non-technical skills usage will be evaluated according to the form developed and published by Cooper et al. (2010) as a Team Emergency Assessment Measure (TEAM) tool based on the Likert scale - Never/Hardly ever (0), Seldom (1), About as often as not (2), Often (3), Always/Nearly always (4).

CONTACTS AND LOCATIONS:
Overall Officials: David Peran, DrPH, Study Chair — Prague Emergency Medical Services; Roman Sykora, PhD, Study Director — Emergency Medical Services of the Karlovy Vary Region; Jana Vidunová, MD, Study Director — Emergency Medical Services of the Pilsner Region; Ivana Krsova, MSc., Principal Investigator — Emergency Medical Services of the Pilsner Region; Jaroslav Pekara, PhD, Principal Investigator — Prague Emergency Medical Services; Patrik C Cmorej, PhD, Principal Investigator — Emergency Medical Services of the Usti nad Labem Region; Nikola Brizgalová, DrPH, Principal Investigator — Emergency Medical Services of the Karlovy Vary Region
Locations (3):
- Czechia (3):
  - Emergency Medical Services of the Karlovy Vary region, Karlovy Vary
  - Emergency Medical Services of the Pilsner region, Pilsen
  - Prague Emergency Medical Services, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper SJ, Cant RP. Measuring non-technical skills of medical emergency teams: an update on the validity and reliability of the Team Emergency Assessment Measure (TEAM). Resuscitation. 2014 Jan;85(1):31-3. doi: 10.1016/j.resuscitation.2013.08.276. Epub 2013 Sep 12. PMID 24036193
- [Background] Napier F, Davies RP, Baldock C, Stevens H, Lockey AS, Bullock I, Perkins GD. Validation for a scoring system of the ALS cardiac arrest simulation test (CASTest). Resuscitation. 2009 Sep;80(9):1034-8. doi: 10.1016/j.resuscitation.2009.04.043. Epub 2009 Jun 13. PMID 19525052
- [Background] PERAN, D., KUBALOVÁ, J..: Observation of non-technical skills during resuscitation (Sledování netechnických dovedností při resuscitaci) [article in Czech language]. Urgentní medicína: Časopis pro neodkladnou lékařskou péči. Mediprax CB s.r.o., 2017 (4). ISSN 1212-1924.
- [Derived] Peran D, Sykora R, Vidunova J, Krsova I, Pekara J, Renza M, Brizgalova N, Cmorej PC. Non-technical skills in pre-hospital care in the Czech Republic: a prospective multicentric observational study (NTS study). BMC Emerg Med. 2022 May 13;22(1):83. doi: 10.1186/s12873-022-00642-4. PMID 35562664